CLINICAL TRIAL: NCT06903845
Title: The Effect of App. for Medication-check and Video-call Guided Education on APIXABAN Adherence in Patients of Atrial Fibrillation With Cardiac Disease: Randomised Control Pilot Study(APIXABAN Study)
Brief Title: APIXABAN App Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dong-Ju Choi (Other)
Responsible Party: Sponsor-Investigator, Dong-Ju Choi, Professor, Seoul National University Bundang Hospital
Organization: Seoul National University Bundang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APIXABAN app
Record Dates: First submitted 2025-03-28; First posted 2025-04-01 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; mobile application; digital health; medication adherence
MeSH Terms: conditions — Atrial Fibrillation; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medication reminder app + video call (Experimental): Patients can use medication reminder app and have video recall
  Interventions: Procedure: video call; Device: Medication reminder app
- Medication reminder app only (Placebo Comparator): Patients can only use medication reminder app and cannot have video recall
  Interventions: Device: Medication reminder app

INTERVENTIONS:
Procedure: video call — Conduct video training every two weeks emphasizing medication adherence.
  Arms: Medication reminder app + video call
Device: Medication reminder app — Medication reminder app will remind patients to take your medication.

SUMMARY:
The aim of this clinical trial is to evaluate whether the medication reminder app and video call can improve medication adherence to apixaban in patients with AF and comorbidities.

Patients with AF and comorbid heart disease taking apixaban who meet the inclusion criteria will be randomised 1:1 to a treatment arm using a medication reminder app and bi-weekly video education and a control arm using the medication reminder app alone to compare medication adherence.

Patients in both groups will use the medication app, but only the treatment group will receive additional education and feedback via video call every two weeks to reinforce the use of the medication app and medication reminders with video education.

The study aims to assess the change in adherence between the two groups at week 8.

ELIGIBILITY:
Participants must meet all of the following criteria:

Adults aged 19 years or older with a diagnosis of atrial fibrillation (AF)

Presence of at least one of the following cardiovascular or metabolic comorbidities:

A. Heart failure

B. Hypertension

C. Coronary artery disease

D. Peripheral arterial disease

E. Diabetes mellitus

F. Stroke

G. Other cardiac diseases requiring treatment

Currently taking or planning to initiate oral anticoagulation therapy with apixaban

Able to use a smartphone with an Android operating system

Voluntarily provided written informed consent to participate in the clinical trial after being adequately informed of its purpose, procedures, and potential risks

2. Exclusion Criteria

Participants will be excluded if any of the following conditions apply:

Creatinine clearance (CCr) < 15 mL/min

Presence of moderate to severe mitral stenosis

History of mitral valve repair or replacement

Clinically significant history of alcohol or substance abuse

Deemed by the investigator to be legally or psychologically unsuitable for participation in the clinical trial

Participation in another clinical trial involving investigational drugs within 4 weeks prior to screening

Declines or is unwilling to provide informed consent for participation in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence by pill count | From enrollment to the end of treatment at 8 weeks
  Medication adherence by pill count: both the value itself and the percentage of 100% achieved

SECONDARY OUTCOMES:
Medication adherence by App. Calculation | From enrollment to the end of treatment at 8 weeks
  Medication adherence by App. Calculation
Clinical composite end poin | From enrollment to the end of treatment at 8 weeks
  Clinical composite end point: including composites of stroke, systemic embolic event, major bleeding requiring hospitalization or transfusion, or death
App adherence by log trail | From enrollment to the end of treatment at 8 weeks
  App adherence by log trail
Change in adherence questionnaire scores from baseline to week 8 | From enrollment to the end of treatment at 8 weeks
  Change in adherence questionnaire scores from baseline to week 8 Rated on a scale of 1 to 5, with higher scores being better

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyeonggido, South Korea

IPD SHARING:
Plan to Share IPD: No